CLINICAL TRIAL: NCT04291248
Title: A Randomized, Open-label , Multi-cohort, Multicenter, Phase II Study of Anlotinib Combined With AK105 Injection in Subjects With MSI-H or dMMR Advanced Solid Tumor
Brief Title: A Study of Anlotinib Combined With AK105 Injection in Subjects With Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Advanced Solid Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AK105-II-03
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2019-12

CONDITIONS: MSI-H or dMMR Advanced Solid Tumors
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib+AK105 injection (Experimental): AK105 200mg intravenously (IV) on day 1 of each 21-day cycle plus Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: AK105; Drug: Anlotinib
- AK105 injection (Experimental): AK105 200mg intravenously (IV) on day 1 of each 21-day cycle.
  Interventions: Drug: AK105

INTERVENTIONS:
Drug: AK105 — AK105 is a humanized monoclonal antibody that specifically binds to PD-1. AK105 has a typical antibody structure and is composed of two lgG1 subtype heavy chains and two kappa subtypes light chains covalently linked by disulfide bonds.
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor.
  Arms: Anlotinib+AK105 injection

SUMMARY:
This study is designed to evaluate the efficacy and safety of Anlotinib combined with AK105 injection or AK105 monotherapy in subjects with MSI-H or dMMR advanced solid tumors. In this study, 138 subjects will be enrolled, and those who met the admission criteria will divide into cohort 1 (anlotinib combined with AK105) and cohort 2 (AK105 ). The first phase of this study is a randomized, open-label, parallel-controlled, multicenter design, in which 30 subjects are randomly enrolled in two cohorts. The second phase is to continue enrollment of cohort 1 or cohort 2 when which cohort has the better clinical benefit than the other one.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathologically confirmed MSI-H or dMMR advanced malignant solid tumors. 2. Has provided previously achieved tumor tissue samples or fresh samples. 3. 18 years and older; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.

  4. At least one measurable lesion. 5. The main organs function are normally. 6.Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

  7.Understood and signed an informed consent form.

Exclusion Criteria:

* 1.Has used against PD-1, PD-L1 and other related immunotherapeutic drugs. 2. Has received chemotherapy, radiotherapy or other treatments within 4 weeks prior to the first dose.

  3. Has brain metastases with symptoms or symptoms control for less than 2 months.

  4. Has diagnosed and/or treated additional malignancy within 3 years prior to the first dose.

  5. Has multiple factors affecting oral medication. 6.Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

  7. Has unrelieved spinal cord compression. 8. Imaging shows that tumors invade large blood vessels. 9. Has hemoptysis within 1 month prior to the first dose and maximum daily hemoptysis ≥2.5 mL.

  10. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  11. Has received surgery, or unhealed wounds within 4 weeks before the first dose.

  12. Has artery/venous thrombosis prior to the first dose within 6 months. 13. Has drug abuse history that unable to abstain from or mental disorders. 14. Has any serious and / or uncontrolled disease. 15. Has received vaccination or attenuated vaccine within 4 weeks prior to the first dose.

  16. Hypersensitivity to recombinant humanized anti-PD-1 monoclonal or its components.

  17. Has active autoimmune diseases requiring systemic treatment occurred within 2 years before the first administration.

  18.Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first dose.

  19. Has a history of active TB. 20. Has participated in other anticancer drug clinical trials within 4 weeks. 20. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by Independent Review Committee (IRC) | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) based on IRC.

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by investigator | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) based on investigator.
Disease control rate（DCR） | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to 96 weeks
  OS defined as the time from the first dose to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences, Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of The PLA Air Force Medical University, Xi’an, Shanxi
  - Shanxi Cancer Hospital, Xi’an, Shanxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality